CLINICAL TRIAL: NCT05793736
Title: A Feasibility Study of an HVR Protocol Biofeedback Training to Manage Long Covid Syndrome Symptoms
Brief Title: Prevention of Long Covid Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Giulia Cossu, Principal Investigator, University of Cagliari
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: NP/2023/496
Record Dates: First submitted 2023-03-21; First posted 2023-03-31 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Post-Acute COVID-19 Syndrome; Biofeedback, Psychology; Quality of Life; Depressive Symptoms; Fatigue; Anxiety; Pain; Cognitive Symptom
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Depression; Fatigue; Anxiety Disorders; Pain; Neurobehavioral Manifestations | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a controlled clinical feasibility trial with three evaluation times (T0 pre-treatment; T1 post treatment five weeks after T0; T2 nine weeks after T1) aimed at verifying the feasibility and tolerability of an intervention performed with biofeedback training (already extensively tested on other clinical populations and free of side effects) and aimed to obtain a preliminary measure of its effectiveness on patients with Long Covid syndrome
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- biofeedback + treatment as usual (Experimental): The selected sample (n 10) will undergo 10 total Biofeedback Training sessions, twice a week. Each session will last 45 minutes. The total duration of the treatment will be 5 weeks, plus standard therapies (treatment as usual)
  Interventions: Device: Biofeedback training
- treatment as usual (Active Comparator): The control sample (n 10) will be treated only with standard therapies (treatment as usual) without the use of biofeedback training
  Interventions: Drug: Treatment as usual

INTERVENTIONS:
Device: Biofeedback training — The intervention lasts 5 weeks, twice a week, each session lasts 45 minutes in which HRV (Heart Rate Variability) is detected, through plethysmographic sensors placed on the finger or earlobe during assigned tasks. During tasks that involve progressively more complex phases, they allow the person to receive immediate feedback on the video screen.
  Arms: biofeedback + treatment as usual
Drug: Treatment as usual — The sample will be treated only with standard therapies (treatment as usual) without the use of biofeedback training
  Arms: treatment as usual

SUMMARY:
Biofeedback equipment is classified by the Food and Drug Administration (FDA) as medical device class II and this type of equipment/treatment has shown evidence regarding stress management in post-Covid-19 syndrome.

The main objective of the study is to verify the feasibility of an HVR biofeedback training protocol in patients with long covid, and also to verify improvement induced by the technique in relation to: cognitive performance; pain perception; fatigue; quality of life; depressive and anxious symptoms

DETAILED DESCRIPTION:
Long COVID is known by different names, and include a wide range of persistent symptoms that develop after SARS-CoV-2 infection and last for usually more than 12 weeks to months and up to 2 years, so far. The most common symptoms categorizable as neurological are fatigue, brain fog, and headache, among respiratory symptoms chest pain and shortness of breath, other less easily classifiable symptoms are heart palpitations and muscle pain. These symptoms are often debilitating enough to leave patients unable to work.

According to the WHO (2023), an estimated 17 million people were thought to be living with the long-term effects of COVID-19. Still now in less active pandemic phases, the risk of developing long COVID symptoms, at 10-20% of those infected, remains just as strong.

Trying to find a solution to manage symptoms through evidence-based practices is considered a current necessity to help health patients and professionals.

Biofeedback allows to learn self-regulation of some physiological processes through feedback of recorded parameters and the goal is improving health and its performances.

Biofeedback measures muscle activity, skin temperature, electrodermal activity (sudoriparous glands activity), respiration, heart rate, blood pressure, electrical brain activity and bloodstream, it also gives a quick feedback of those personal measurements to the patient, in this way biofeedback teaches people to have a more active role in maintaining a good personal, mental and physical health (quickly and thoroughly it give person feedback of activity and biofeedback teaches people to take a more active role in maintaining personal health and mental health and physical health).

Biofeedback equipment is classified by the Food and Drug Administration (FDA) as medical device class II and this type of equipment/treatment has shown evidence regarding stress management (evidence were shown as regards stress menagement).

The greatest benefits from using biofeedback are: improvement of sleep quality, improvement of self- efficacy, improvement of pain threshold, and improvement of emotional adjustment. In particular, a study conducted with HRV biofeedback, in which the sample learned resonance frequency breathing, showed dicreases in depression and pain and improved the person's system functioning.

Study objectives

The main objective of the study is to verify the feasibility of an HVR biofeedback training protocol in patients with Long Covid syndrome, and also to produce a preliminary measurement of the possible improvement induced by the technique in relation to:cognitive performance; pain perception; fatigue; quality of life; depressive and anxious symptoms. This measure will be useful to estimate the expected improvement in future case-control studies. Study design

This is a controlled clinical trial between usual care and biofeedback training plus usual care.

ELIGIBILITY:
Inclusion Criteria:

* People who have contracted Covid-19 and have symptoms attributable to Long syndrome

Exclusion Criteria:

* patients with cognitive difficulties and/or diagnosis of mental retardation
* patients with severe comorbidities with the exception of anxious/depression symptoms arising in conjunction with the viral infection or long covid syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 5 weeks and to 9 weeks in Patient Health Questionnaire-9 (PHQ-9) score | T0 (0 weeks); T1 (5weeks); T2 (9 weeks)
  short self-administered tool used for screening, diagnosis, monitoring and measuring the severity of depression. It's composed of 9 items that correspond to the symptoms of major depression according to DSM-IV. The score has a range between 0 and 27. Scores between 0 and 9 indicate the presence of a sub-threshold depression. The score of 10 is indicated as the point at which the sensitivity and specificity of the instrument are recognized as optimal for highlighting depressions of clinical relevance
Change from Baseline to 5 weeks and to 9 weeks in Brief Fatigue Inventory (BFI) score | T0 (0 weeks); T1 (5weeks); T2 (9 weeks)
  The Brief Fatigue Inventory (BFI) is a brief screening tool designed to assess the severity and impact of fatigue on daily functioning.
Change from Baseline to 5 weeks and to 9 weeks in Short Form Health Survey (SF-12) score | T0 (0 weeks); T1 (5weeks); T2 (9 weeks)
  The Short Form Health Survey (SF-12), brief version of SF-36 questionnaire, made up of twelve questions, includes the following dimensions: physical activity, disturbance in physical health, physical condition, self-assessment of health status, vitality, social activity and mental health. Higher SF-12 scores recorded a greeting and QoL performance.
Change from Baseline to 5 weeks and to 9 weeks in Matrix test (Spinnler H, Tognoni G., 1987) score | T0 (0 weeks); T1 (5weeks); T2 (9 weeks)
  Evaluates the indicators of selective attention
Change from Baseline to 5 weeks and to 9 weeks in Trail Making Test (Giovagnoli et al.,1996) score | T0 (0 weeks); T1 (5weeks); T2 (9 weeks)
  Evaluates cognitive functions such as cognitive flexibility and inhibitory control and attention
Change from Baseline to 5 weeks and to 9 weeks in Digit Span (Orsini et al., 1987; Mondini et al., 2003) score | T0 (0 weeks); T1 (5weeks); T2 (9 weeks)
  Evaluate verbal short-term memory and working memory
Change from Baseline to 5 weeks and to 9 weeks in Stroop Test (Caffarra et al.; 2002) score | T0 (0 weeks); T1 (5weeks); T2 (9 weeks)
  Evaluates selective attention, the processes of inhibition of irrelevant information and cognitive flexibility
Change from Baseline to 5 weeks and to 9 weeks in Frontal Assessment Battery - FAB (Dubois et al.; 2000) score | T0 (0 weeks); T1 (5weeks); T2 (9 weeks)
  It is a functionality screening battery global executive performance by means of a series of cognitive and behavioral tests
Change from Baseline to 5 weeks and to 9 weeks in Rey's Word Test (Caltagirone et al. 1995) score | T0 (0 weeks); T1 (5weeks); T2 (9 weeks)
  Evaluates long-term memory, semantic memory, specifies in which phase of the mnemonic process the deficit is
Change in Checklist on tolerability, possible side effects after the biofeedback session | At the end of each biofeedback session
  Checklist on tolerability, possible side effects after the biofeedback session
Intervention satisfaction questionnaire | T1 (5weeks)
  Intervention satisfaction questionnaire
Change from Baseline to 5 weeks and to 9 weeks in Visual Analog Scale VAS (Scott Huskisson, 1976) score | T0 (0 weeks); T1 (5weeks); T2 (9 weeks)
  Allows you to have a visual representation of the amplitude of the pain perceived by the person ache
Change from Baseline to 5 weeks and to 9 weeks in Self-Rating Anxiety Scale (SAS) score | T0 (0 weeks); T1 (5weeks); T2 (9 weeks)
  SAS is a 20-item self-report assessment device built to measure anxiety levels, based on scoring in 4 groups of manifestations: cognitive, autonomic, motor and central nervous system symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- P.O. San Giovanni di Dio, AOU Cagliari, Cagliari, Italy